CLINICAL TRIAL: NCT01327079
Title: Optimizing the Use of Methadone in Newborn Infants
Brief Title: The Use of Methadone in Newborn Infants
Acronym: Methadone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John van den Anker (Other)
Responsible Party: Sponsor-Investigator, John van den Anker, John van denanker, MD, PhD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4781; IV Methadone (Other Grant/Funding Number: KDA027992A)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Premature Birth of Newborn; Critically Ill
Keywords: NICU; Methadone; neonates
MeSH Terms: conditions — Premature Birth; Critical Illness | interventions — Methadone; Inulin; sinistrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Gestational age less than 29 weeks We will substitute for one study dose 0.1 mg morphine with 0.1 mg methadone, whereas if the infant has been treated with fentanyl substitute for that one study dose 1 μg fentanyl with 0.1 mg methadone.
  Administration of inulin:
  Inulin will be administered as a glucose 10%-inulin solution containing 25 gr. inulin/L, at an infusion rate of 0.6 mL/kg/h. After 24 h, the inulin clearance will be calculated.
  Interventions: Drug: Methadone
- Group 2 (Experimental): Gestational age greater then 29 weeks We will substitute for that one study dose 0.1 mg morphine with 0.1 mg methadone, whereas if the infant has been treated with fentanyl substitute for that one study dose 1 μg fentanyl with 0.1 mg methadone.
  Administration of inulin:
  Inulin will be administered as a glucose 10%-inulin solution containing 25 gr. inulin/L, at an infusion rate of 0.6 mL/kg/h. After 24 h, the inulin clearance will be calculated.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — If the infant has been treated with morphine than substitute for that one study dose 0.1 mg morphine with 0.1 mg methadone, whereas if the infant has been treated with fentanyl substitute for that one study dose 1 μg fentanyl with 0.1 mg methadone.
  Administration of inulin:
  Inulin will be administered as a glucose 10%-inulin solution containing 25 gr. inulin/L, at an infusion rate of 0.6 mL/kg/h. After 24 h, the inulin clearance will be calculated.
  Other Names: inulin
  Arms: Group 1
Drug: Methadone — If the infant has been treated with morphine than substitute for that one study dose 0.1 mg morphine with 0.1 mg methadone, whereas if the infant has been treated with fentanyl substitute for that one study dose 1 μg fentanyl with 0.1 mg methadone.
  Administration of inulin:
  Inulin will be administered as a glucose 10%-inulin solution containing 25 gr. inulin/L, at an infusion rate of 0.6 mL/kg/h. After 24 h, the inulin clearance will be calculated.
  Other Names: inulin (Sinistrin)

SUMMARY:
This proposed investigation will test the following hypotheses: 1) Enzymatic activity of CYP2B6 characterized by the formation clearance of methadone to EDDP (CLf,EDDP), is directly related to both gestational and postnatal age; 2) variations in the CYP2B6 gene (SNPs) are associated with variable activity of the CYP2B6 enzyme (as measured by the formation clearance, CLf,EDDP), and 3) the elimination rate of methadone and its major metabolite EDDP in neonates is dependent on the glomerular filtration rate and therefore on the stage of development (defined by both gestational and postnatal age). The investigators propose to develop a PK model for methadone dosing in neonates that takes into account both developmental stage and genetic variability. The long-term goal of the proposed investigations is to improve dosing of methadone in neonates exposed to opioids in utero or post-natally, leading to improved control of their withdrawal syndrome and decreased adverse drug reactions associated with the current use of methadone in these vulnerable patients. More immediately, the investigators will develop a PK model for methadone dosing based on relevant developmental and genetic characteristics. The acquired knowledge based on the proposed study will lead to a more efficacious treatment of pain or opiate withdrawal syndrome in newborn infants with a decreased chance of adverse drug reactions.

DETAILED DESCRIPTION:
The investigators will identify and recruit from the NICU of CNMC 60 preterm neonates uniformly distributed with respect to gestational age and encompassing GA's of from 22 to less than 43 weeks.

* Stratified Selection by Gestational Age (GA): The study neonates will be selected to achieve balance in the following GA strata: (22-24 wks, 25-26 wks, 27-28 wks, 29-30 wks, 31-32 wks, 33-37 wks; 38-43 wks). Stratification will be done to ensure broad representation by GA. As described below, analyses will treat GA as a continuous variable.
* Randomization will assign a newborn infant to group 1 (n=30) or group 2 (n=30).
* Study medications: Methadone and inulin administration Blood and urine will be collected for the purposes of this research project. Blood will be drawn from the indwelling arterial catheter that already is in place for clinical purposes. The amount of blood obtained for all study related determinations will be minimized and kept at less than 3 mL/kg of blood per 48 hour period. The study will last 60 hours for group 1 and 72 hours for group.
* DNA study 0.3ml whole blood will be collected from each subject
* PK study Blood samples (0.2 mL per sample) will be taken in 30 newborn infants at t=0, 1, 4, 12, 36, 60 h (group 1) after the administration of one dose of methadone, and in 30 newborn infants at t=0, 2, 8, 24, 48, 72 hr (group 2) after the administration of methadone. A total of 1.5 ml of blood will be collected from each subject
* Urine Collection Urine samples will be collected from each infant's diaper (wood pulp based study diapers) every 3-4 hours over the first 24 hour period or alternatively, from an indwelling urinary catheter placed based on clinical indications unrelated to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants of both genders and all races who have:

  * a postnatal age of less than 3 months
  * an indwelling (peripheral or umbilical) arterial line, and
  * already treated with an opioid (morphine or fentanyl) for clinical reasons

Exclusion Criteria:

* Neonates with severe asphyxia grade III or IV intraventricular hemorrhage,
* Neonates with major congenital malformations or facial malformations (e.g., cleft lip and palate), neurological disorders
* Neonates receiving continuous or intermittent neuromuscular blockers neonates will be excluded who have:

  * clinical or biochemical evidence of hepatic and renal failure (including systemic hypoperfusion
  * received drugs that are CYP2B6 substrates
  * been exposed in utero to methadone, despite the fact that they indeed receive a CYP2B6 substrate through their mother, will not be excluded but will be analyzed as a subgroup

Ages: 22 Weeks to 43 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Methadone PK and EDDP | 36 months
  Primary outcome: Plasma and urine levels of methadone and EDDP (2-ethylidene- 1,5-dimethyl-3,3-diphenylpyrrolidine, the main metabolite of methadone). Secondary endpoints: CYP2DB6 genetic variability.

SECONDARY OUTCOMES:
DNA | 36 months
  Secondary endpoints: CYP2DB6 genetic variability.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens Research Institute, Washington D.C., District of Columbia
  - Childrens's Research Institute, Washington D.C., District of Columbia

REFERENCES:
- [Derived] van Donge T, Samiee-Zafarghandy S, Pfister M, Koch G, Kalani M, Bordbar A, van den Anker J. Methadone dosing strategies in preterm neonates can be simplified. Br J Clin Pharmacol. 2019 Jun;85(6):1348-1356. doi: 10.1111/bcp.13906. Epub 2019 Apr 10. PMID 30805946